CLINICAL TRIAL: NCT02204657
Title: The Effect of Professional Continuous Glucose Monitoring on Diabetes Management,Hypoglycemia and Glycemic Control in Insulin-requiring Gestational Diabetes Mellitus
Brief Title: The Effect of Continuous Glucose Monitoring on Glycemic Control in Insulin-requiring Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Shireene Vethakkan, Associate Professor and Consultant Endocrinologist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 961.7; PPUM/QSU/300-04/11 (Other: University Malaya Medical Centre, Malaysia)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-06

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Continuous glucose monitoring in GDM
MeSH Terms: conditions — Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Glucose Monitoring System (Active Comparator): Patients in this arm will receive Continuous Glucose Monitoring System (CGMS) at 28,32 and 36 weeks of gestation and their insulin titrated according to the CGMS results.
  Interventions: Device: Continuous Glucose Monitoring System
- Control (No Intervention): Patients in this arm will not receive any Continuous Glucose Monitoring System( CGMS) and the insulin titration will be made based on their fingerstick sugar readings.

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — Patients in the intervention group will receive Continuous Glucose Monitoring(CGMS) at weeks 28, 32 and 36 and have the CGMS reviewed at weeks 29, 33 and 37 and management adjusted based on the CGMS readings
  Other Names: iPro, Medtronic
  Arms: Continuous Glucose Monitoring System

SUMMARY:
The purpose of this study is to determine if professional Continuous glucose monitoring improves glycemic control with less hypoglycaemia in insulin-requiring Gestational Diabetes Mellitus

DETAILED DESCRIPTION:
1. OBJECTIVES

   1. To determine if professional CGM improves glycemic control with less hypoglycaemia in insulin- requiring GDM
   2. To determine if professional CGM use alters management of insulin-requiring GDM
   3. To determine if professional CGM improves pregnancy outcomes in insulin-requiring GDM.
   4. To determine patient attitudes toward CGMS.
2. HYPOTHESES

   1. Professional CGMS improves glycaemic control in women with insulin-requiring GDM with less hypoglycaemia
   2. Professional CGM use will alter management of insulin-requiring GDM
   3. Professional CGMS will reduce perinatal morbidity and mortality in patients with insulin- requiring GDM
   4. Third trimester CGMS parameters will correlate better with perinatal outcomes compared with conventional measures of glycaemic control in pregnancy i.e. fructosamine/ A1c/ FBS/ 2hrs PP glucose

STUDY DESIGN

* This is a prospective, open-label, randomized controlled trial. We plan to recruit 80 women with gestational diabetes at 28 weeks gestation or less from the UMMC antenatal clinic. These women should be insulin-naïve but require insulin therapy. 40 subjects (Group 1) will be selected to undergo professional CGM at weeks 28, 32, and week 36 and another 40 subjects individually matched with regards, to age, baseline A1c, BMI will be recruited to undergo usual antenatal care without CGMS (Group 2). The CGMS data will be uploaded and reviewed at weeks 29, 33, and 37 and changes made to the therapeutic regimen as required by the endocrinologist. All mothers will be required to measure their glucose levels at 7 standardized points in a day daily. These glucose readings will be recorded in a diary together with a food log. All subjects will also be required to keep a hypoglycaemia diary.
* The primary outcomes will be glycaemic control in the third trimester and maternal hypoglycaemia. We also plan to assess changes to management made by the endocrinologist based on the additional information on glycemic control obtained from professional CGM use. We also plan to compare hypoglycaemia and hyperglycaemia detection rates using the CGMS and fingerstick methods of glucose evaluation. Patient satisfaction in both groups will also be assessed. Written and informed consent will be obtained in accordance with the principles of the Helsinki Declaration

ELIGIBILITY:
Inclusion Criteria:

* women with gestational diabetes
* aged >18 years
* less than or equal to 28 weeks gestation of pregnancy
* singleton pregnancy
* insulin naive , but requiring insulin therapy

Exclusion Criteria:

* pregestational type 1 or 2 diabetes mellitus
* newly diagnosed overt diabetes in pregnancy ( HbA1c > 6.5)
* hypothyroidism
* Cushing's syndrome/ using exogenous steroids
* chronic infection ( HIV, Hepatitis B/C, Tuberculosis)
* any active chronic systemic disease ( except essential hypertension)
* assisted conception
* pregnancies with fetal anomalies / where imminent or preterm delivery is likely because of maternal disease ( besides gestational diabetes)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shireene R Vethakkan, MBBS,MD, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy HR, Rayman G, Lewis K, Kelly S, Johal B, Duffield K, Fowler D, Campbell PJ, Temple RC. Effectiveness of continuous glucose monitoring in pregnant women with diabetes: randomised clinical trial. BMJ. 2008 Sep 25;337:a1680. doi: 10.1136/bmj.a1680. PMID 18818254
- [Background] Chen R, Yogev Y, Ben-Haroush A, Jovanovic L, Hod M, Phillip M. Continuous glucose monitoring for the evaluation and improved control of gestational diabetes mellitus. J Matern Fetal Neonatal Med. 2003 Oct;14(4):256-60. doi: 10.1080/jmf.14.4.256.260. PMID 14738172
- [Background] Yogev Y, Visser GH. Obesity, gestational diabetes and pregnancy outcome. Semin Fetal Neonatal Med. 2009 Apr;14(2):77-84. doi: 10.1016/j.siny.2008.09.002. Epub 2008 Oct 15. PMID 18926784
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Tan PC, Ling LP, Omar SZ. The 50-g glucose challenge test and pregnancy outcome in a multiethnic Asian population at high risk for gestational diabetes. Int J Gynaecol Obstet. 2009 Apr;105(1):50-5. doi: 10.1016/j.ijgo.2008.11.038. Epub 2009 Jan 19. PMID 19154997
- [Background] Balaji V, Balaji M, Anjalakshi C, Cynthia A, Arthi T, Seshiah V. Inadequacy of fasting plasma glucose to diagnose gestational diabetes mellitus in Asian Indian women. Diabetes Res Clin Pract. 2011 Oct;94(1):e21-3. doi: 10.1016/j.diabres.2011.07.008. Epub 2011 Aug 10. PMID 21831468
- [Background] Klonoff DC, Buckingham B, Christiansen JS, Montori VM, Tamborlane WV, Vigersky RA, Wolpert H; Endocrine Society. Continuous glucose monitoring: an Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2011 Oct;96(10):2968-79. doi: 10.1210/jc.2010-2756. PMID 21976745
- [Background] Klonoff DC. Continuous glucose monitoring: roadmap for 21st century diabetes therapy. Diabetes Care. 2005 May;28(5):1231-9. doi: 10.2337/diacare.28.5.1231. No abstract available. PMID 15855600
- [Background] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Lain KY, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A multicenter, randomized trial of treatment for mild gestational diabetes. N Engl J Med. 2009 Oct 1;361(14):1339-48. doi: 10.1056/NEJMoa0902430. PMID 19797280
- [Background] Sathyapalan T, Mellor D, Atkin SL. Obesity and gestational diabetes. Semin Fetal Neonatal Med. 2010 Apr;15(2):89-93. doi: 10.1016/j.siny.2009.09.002. Epub 2009 Oct 28. PMID 19875346
- [Derived] Paramasivam SS, Chinna K, Singh AKK, Ratnasingam J, Ibrahim L, Lim LL, Tan ATB, Chan SP, Tan PC, Omar SZ, Bilous RW, Vethakkan SR. Continuous glucose monitoring results in lower HbA1c in Malaysian women with insulin-treated gestational diabetes: a randomized controlled trial. Diabet Med. 2018 Aug;35(8):1118-1129. doi: 10.1111/dme.13649. Epub 2018 May 23. PMID 29663517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 women with insulin-requiring gestational diabetes enrolled from the University of Malaya Medical CentreAntenatal Clinic between April 2013 to April 2015.
  Women with overt diabetes or pregestational diabetes were excluded.
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring System | Control
Started | 32 | 25
Completed | 25 | 25
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitoring System | Control | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.80 (4.53) | 32.6 (4.93) | 32.7 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malaysia | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control by Measurement of HbA1c
Time Frame: From 28 weeks until delivery
Measure: Mean (Standard Deviation); unit: mean percentage
Arm/Group | Continuous Glucose Monitoring System | Control
Number analyzed (Participants) | 25 | 25
mean percentage | 5.17 (0.41) | 5.57 (0.57)

2. Secondary Outcome: Hypoglycemia
Time Frame: 28 weeks until delivery
Measure: Median (Inter-Quartile Range); unit: episodes per patient
Arm/Group | Continuous Glucose Monitoring System | Control
Number analyzed (Participants) | 25 | 25
episodes per patient | 8.0 [3 to 14] | 4.0 [1 to 6.5]

ADVERSE EVENTS:
Arm/Group | Continuous Glucose Monitoring System | Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No